CLINICAL TRIAL: NCT02556983
Title: Optimizing the Radiation Dose for CT Imaging With Iterative Reconstruction in Diagnosing Acute Appendicitis: Dose Simulation Study
Brief Title: CT Dose Simulation Study for Appendicitis
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ji Hoon Park, Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: SNUBH-02-2015-030
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Appendicitis
Keywords: Appendicitis; Tomography, X-Ray Computed; Receiver operating characteristic (ROC) Curve; Computer Simulation
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected appendicitis: Patients who are suspected as having acute appendicitis
  Interventions: Radiation: CT

INTERVENTIONS:
Radiation: CT — Contrast-enhanced CT images of the abdomen and pelvis will be obtained during the portal venous phase using a 256-channel CT system (Philips Healthcare, Cleveland, OH). The target median dose-length product (DLP) is 130 mGy·cm, which corresponded to an effective dose of 2 mSv with a conversion factor of 0.015 mSv·mGy-1·cm-1. The radiation output was automatically adjusted according to the individual patient's body size.

SUMMARY:
The study will explore CT radiation dose as low as reasonably achievable in diagnosing acute appendicitis, by using of dose simulation technique and iterative reconstruction.

DETAILED DESCRIPTION:
Three sequential non-inferiority tests are planned. First, three readers will review the original 2-mSv images. Second, the readers will review the 75%-dose images. After the readers review the 75%-dose images and before the readers reviewed the 50%-dose images, the non-inferiority of 75% dose to the original dose will be tested. If the non-inferiority is not accepted, the study will be terminated with the conclusion of 2 mSv as the lowest acceptable dose. If the non-inferiority is accepted, the study will be continue to the next step. In the same manner, the readers will review the next lower-dose images (50% and then 25%), and then the noninferiority will be tested against the original dose.

ELIGIBILITY:
Inclusion Criteria:

* 18-44 years of age.
* Emergency department visit with suspected symptoms and signs of acute appendicitis
* Intravenous contrast-enhanced computed tomography examination requested due to suspicion of appendicitis

Exclusion Criteria:

* having contraindications of intravenous contrast agent

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Emergency department visit with suspected symptoms and signs of acute appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance at original dose (2 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 2 months
  The pooled area under curve (AUC) from three radiologists
Diagnostic performance at 75% dose (1.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 1 months
  The pooled AUC from three radiologists
Diagnostic performance at 50% dose (1.0 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 8 months
  *The analysis of 50%-dose CT images will be performed only if non-inferiority of 75%-dose CT to the original CT is proven in terms of the pooled AUC.
  The pooled AUC from three radiologists
Diagnostic performance at 25% dose (0.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 14 months
  *The analysis of 25%-dose CT images will be performed only if non-inferiority of 50%-dose CT is proven to the original CT in terms of the pooled AUC.
  The pooled AUC from three radiologists

SECONDARY OUTCOMES:
Sensitivity at original dose (2 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 2 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Specificity at original dose (2 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 2 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Sensitivity at 75% dose (1.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 1 month
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Specificity at 75% dose (1.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 1 month
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Sensitivity at 50% dose (1.0 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 8 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Specificity at 50% dose (1.0 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 8 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Sensitivity at 25% dose (0.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 14 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Specificity at 25% dose (0.5 mSv) using 5-grade Likert score for the likelihood of appendicitis assigned by each radiologist | 14 months
  For calculation of sensitivity and specificity, the 5-grade scores are collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
Diagnostic confidence in diagnosing and ruling out appendicitis at original CT: the likelihood score for appendicitis | 2 months
  Likelihood score for appendicitis in patients confirmed as having appendicitis Likelihood score for appendicitis in patients confirmed as not having appendicitis
Diagnostic confidence in diagnosing and ruling out appendicitis at 75%-dose CT: the likelihood score for appendicitis | 1 month
  Likelihood score for appendicitis in patients confirmed as having appendicitis Likelihood score for appendicitis in patients confirmed as not having appendicitis
Diagnostic confidence in diagnosing and ruling out appendicitis at 50%-dose CT: the likelihood score for appendicitis | 8 month
  Likelihood score for appendicitis in patients confirmed as having appendicitis Likelihood score for appendicitis in patients confirmed as not having appendicitis
Diagnostic confidence in diagnosing and ruling out appendicitis at 25%-dose CT: the likelihood score for appendicitis | 14 month
  Likelihood score for appendicitis in patients confirmed as having appendicitis Likelihood score for appendicitis in patients confirmed as not having appendicitis
Diagnostic confidence in diagnosing and ruling out appendicitis at original CT: normal appendix visualization rate | 2 month
  The frequency of normal appendix visualization at CT
Diagnostic confidence in diagnosing and ruling out appendicitis at 75%-dose CT: normal appendix visualization rate | 1 month
  The frequency of normal appendix visualization at CT
Diagnostic confidence in diagnosing and ruling out appendicitis at 50%-dose CT: normal appendix visualization rate | 8 months
  The frequency of normal appendix visualization at CT
Diagnostic confidence in diagnosing and ruling out appendicitis at 25%-dose CT: normal appendix visualization rate | 14 months
  The frequency of normal appendix visualization at CT
Diagnostic confidence in diagnosing and ruling out appendicitis at original CT: indeterminate CT interpretation | 2 months
  The frequency of indeterminate CT interpretation (grade 3)
Diagnostic confidence in diagnosing and ruling out appendicitis at 75%-dose CT: indeterminate CT interpretation | 1 month
  The frequency of indeterminate CT interpretation (grade 3)
Diagnostic confidence in diagnosing and ruling out appendicitis at 50%-dose CT: indeterminate CT interpretation | 8 months
  The frequency of indeterminate CT interpretation (grade 3)
Diagnostic confidence in diagnosing and ruling out appendicitis at 25%-dose CT: indeterminate CT interpretation | 14 months
  The frequency of indeterminate CT interpretation (grade 3)
Alternative diagnoses at original CT: the radiologists will record possible alternative diagnosis if the patients are presumed to be not having appendicitis | 2 months
  The numbers of important alternative diagnoses established
Alternative diagnoses at 75%-dose CT: the radiologists will record possible alternative diagnosis if the patients are presumed to be not having appendicitis | 1 month
  The numbers of important alternative diagnoses established
Alternative diagnoses at 50%-dose CT: the radiologists will record possible alternative diagnosis if the patients are presumed to be not having appendicitis | 8 months
  The numbers of important alternative diagnoses established
Alternative diagnoses at 25%-dose CT: the radiologists will record possible alternative diagnosis if the patients are presumed to be not having appendicitis | 14 months
  The numbers of important alternative diagnoses established

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Park, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bunadang Hospital, Seongnam-si, Gyeonggi-do, South Korea